CLINICAL TRIAL: NCT05769127
Title: Baltimore Metropolitan Diabetes Regional Partnership (BMDRP) Diabetes Prevention Program and Diabetes Self-Management Training Outcomes
Brief Title: Diabetes Prevention and Education
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding withdrawn
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, KASHIF M MUNIR, Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HP-00102730
Record Dates: First submitted 2023-02-22; First posted 2023-03-15 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Diabetes; Pre Diabetes; Fatty Liver; Body Weight Changes
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Fatty Liver; Body Weight Changes | interventions — dentin sialophosphoprotein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All subjects participating in the diabetes prevention program will be offered body composition analysis and liver fat analysis, before, during, and after the lifestyle intervention
  Interventions: Other: Diabetes Prevention Program (DPP), Diabetes Self-Management Training (DSMT)

INTERVENTIONS:
Other: Diabetes Prevention Program (DPP), Diabetes Self-Management Training (DSMT) — DPP lifestyle intervention program DSMT education on diabetes and lifestyle changes

SUMMARY:
Type 2 diabetes mellitus is one of the fastest growing public health problems in developed and developing countries and imposes a large financial burden on health-care systems. Preventing, delaying, and managing diabetes should be a priority for health-care systems. Nationally, 38% of adults have prediabetes, with more than 80% of people with prediabetes being unaware of their condition. In Maryland, an estimated 10.5% of adults report prediabetes, and 33.7% of Baltimore City residents have obesity, an important risk factor for prediabetes.

The BMDRP aims to increase the capacity of BMDRP hospitals and community partners to offer DPP and DSMT directly in communities and will also increase the number of referrals into these programs.

Successful enrollment and completion of DPP has demonstrated reduced risk of developing type 2 diabetes for individuals with pre-diabetes. However, limited data exist on changes in body composition and liver fat in individuals completing DPP. Individuals with pre-diabetes often have obesity and non-alcoholic fatty liver disease. We will evaluate for changes in body fat and liver fat in individuals completing the DPP program.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is one of the fastest growing public health problems in developed and developing countries and imposes a large financial burden on health-care systems. Preventing, delaying, and managing diabetes should be a priority for health-care systems. Nationally, 38% of adults have prediabetes, with more than 80% of people with prediabetes being unaware of their condition. In Maryland, an estimated 10.5% of adults report prediabetes, and 33.7% of Baltimore City residents have obesity, an important risk factor for prediabetes. There is racial disparity in obesity prevalence in the City, with obesity prevalence at 22.2% among White, Non-Hispanic adults and 42.0% among Black, Non-Hispanic adults. Several randomized controlled trials have successfully proven that an intensive lifestyle intervention, like the one studied in the Diabetes Prevention Program, can delay the onset of the progression from prediabetes to type 2 diabetes. These studies have shown a decrease in relative risk of type 2 diabetes up to 60% by intensive lifestyle interventions. The National Diabetes Prevention Program is a CDC-recognized yearlong lifestyle change program that is based on these successful trials.

Type 2 diabetes is the leading cause of blindness, lower extremity amputations, and kidney disease requiring dialysis. Diabetes and its complications are primary or secondary factors in an estimated 9 percent of hospitalizations. According to the data from Maryland Behavioral Risk Factor Surveillance System (BRFSS), 14.4% of Baltimore City adult residents and 26.9% of residents aged 65 and older have diabetes, compared to 12.1% of adults statewide. The goals of Diabetes Self-Management Training (DSMT) are to improve glycemic control and reduce the risk of micro and macro-vascular complications as supported by numerous epidemiologic and interventional studies.

Health inequities are present across the Baltimore Metropolitan region. In Baltimore City, mortality rates from diabetes are almost twice as high for Black residents than for White residents (44.5 vs 23.8 deaths per 100,000 population). The BMDRP aims to increase the capacity of BMDRP hospitals and community partners to offer DPP and DSMT directly in communities and will also increase the number of referrals into these programs. Wrap-around services are critical elements of the BMDRP to mitigate the effects of poverty, food insecurity, and transportation barriers. These services will support the success of individuals in the target population and their ability to achieve diabetes prevention and management goals which will support improved health outcomes.

Successful enrollment and completion of DPP has demonstrated reduced risk of developing type 2 diabetes for individuals with pre-diabetes. However, limited data exist on changes in body composition and liver fat in individuals completing DPP. Individuals with pre-diabetes often have obesity and non-alcoholic fatty liver disease. We will evaluate for changes in body fat and liver fat in individuals completing the DPP program.

ELIGIBILITY:
Inclusion Criteria:

* Qualify for DPP with a diagnosis of pre-diabetes and elevated BMI (≥25 kg/m2 , ≥23kg/m2 if Asian)
* For DSMT, individuals with type 2 diabetes

Exclusion Criteria:

- Normoglycemia

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Enrollees into DPP and DSMT | end of calendar year enrollment, yearly for 3 years
  Measure enrolled participants in DPP or DSMT programs
Change in body weight for DPP participants | 12 months
  Change in weight from baseline to 12 months after participating in DPP lifestyle intervention

SECONDARY OUTCOMES:
Change in diabetes control for DSMT participants | 12 months
  Change in hemoglobin A1c from baseline to 12 months after enrolling in diabetes education program
change in body composition in DPP participants | 12 months
  change in body fat and lean body mass from baseline to 12 months after completing DPP lifestyle intervention (body fat in %, with lower body fat % better outcome)
change in liver elastography in DPP participants | 12 months
  change in liver fat and stiffness assessed by Fibroscan at baseline and 12 months after DPP lifestyle intervention (lower liver fat and stiffness better outcomes)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Center for Diabetes and Endocrinology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No